CLINICAL TRIAL: NCT00763347
Title: A Phase 2, Double-Blind Randomized, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate Treatment With SYR-619 in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety Study of SYR-619 in Treating Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntarily terminated based on preliminary non-clinical findings.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-SYR-619-003; U1111-1124-2377 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SYR-619 12.5 mg QD (Experimental)
  Interventions: Drug: SYR-619
- SYR-619 50 mg QD (Experimental)
  Interventions: Drug: SYR-619
- SYR-619 100 mg QD (Experimental)
  Interventions: Drug: SYR-619
- SYR-619 200 mg QD (Experimental)
  Interventions: Drug: SYR-619
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Alogliptin 25 mg QD (Active Comparator)
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: SYR-619 — SYR-619 12.5 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: SYR-619 12.5 mg QD
Drug: SYR-619 — SYR-619 50 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: SYR-619 50 mg QD
Drug: SYR-619 — SYR-619 100 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: SYR-619 100 mg QD
Drug: SYR-619 — SYR-619 200 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: SYR-619 200 mg QD
Drug: Placebo — SYR-619 placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: SYR-322
  Arms: Alogliptin 25 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of SYR-619, once daily (QD), in subjects with type 2 diabetes mellitus who have not achieved glycemic control with diet and exercise, or by taking metformin.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% is type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected, placing an ever increasing burden on families and the health care system.

SYR-619 is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the in vivo degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide.

The aim of this study is to evaluate the dose-response efficacy, safety and tolerability of treatment with SYR-619 in subjects with type 2 diabetes who do not previously achieve adequate glycemic control with lifestyle modification (diet/exercise) or metformin or sulfonylurea oral antidiabetic monotherapy.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 14 Weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs including sitting and standing blood pressure and pulse, body height and weight, physical examinations, electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with a historical diagnosis of type 2 diabetes mellitus.
* Treatment for diabetes with either lifestyle modification or metformin or sulfonylurea alone for at least the 2 months prior to Screening; and a stable dose of either metformin or sulfonylurea for at least 12 weeks prior to randomization for subjects receiving metformin or sulfonylurea at Screening.
* Those subjects receiving metformin or sulfonylurea monotherapy at randomization must have been at least 75% compliant with their metformin or sulfonylurea regimen during the run in/stabilization period, as assessed by subject diary and investigator assessment.
* No treatment with antidiabetic agents other than metformin alone or sulfonylurea alone within the 3 months prior to Screening.
* Glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive, and a fasting plasma glucose <275 mg/dL (<15.27 mmol/L) at the Week -1 visit.
* Body mass index ≥23 and ≤45 kg/m2.
* Fasting C-peptide concentration ≥0.8 ng/mL (≥0.26 nmol/L). (If this screening criterion is not met, the subject still qualifies if C-peptide ≥1.5 ng/mL [≥0.50 nmol/L] after a challenge test).
* If regular use of other non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
* Systolic blood pressure <160 mm Hg and diastolic pressure <100 mm Hg.
* Hemoglobin ≥12 g/dL (≥120 gm/L) for males and ≥10 g/dL (≥100 gm/L) for females.
* Alanine aminotransferase ≤3 x upper limit of normal.
* Serum creatinine <1.5 mg/dL (<133 micromol/L) for males and <1.4 mg/dL (<124 micromol/L) for females.
* Urine albumin/creatinine ratio of <1000 μg/mg (113 mg/mol) at Screening. If elevated, the subject may be rescreened within 1 week.
* Thyroid-stimulating hormone level ≤ the upper limit of the normal range and the subject has normal thyroid function (clinically euthyroid)
* A female subject of childbearing potential who is sexually active must agree to use adequate contraception, and must be neither pregnant nor lactating from Screening and throughout the duration of the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the subject from completing the study.

Exclusion Criteria:

* Concurrently treated with combined metformin and sulfonylurea antidiabetic therapy.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening.
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* History of treated diabetic gastric paresis.
* New York Heart Association Class III or IV heart failure regardless of therapy.
* Currently treated subjects who are stable at Class I or II are candidates for the study.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that in the investigator's opinion will affect the subject's ability to participate in the study.
* History of alcohol abuse or substance abuse within the 2 years prior to Screening.
* The subject is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Treatment with antidiabetic agents other than study drug or metformin or sulfonylurea is not allowed within the 3 months prior to Screening and through the completion of the end-of-treatment/early termination procedures.
  * Treatment with weight-loss drugs, any investigational antidiabetic drugs, or oral or systemically injected glucocorticoids is not allowed from 3 months prior to randomization through the completion of the end-of-treatment/early termination procedures.
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening.
* Prior treatment in an investigational study of SYR-619 or alogliptin.
* The subject has a known hypersensitivity to any compound related to SYR-619 or alogliptin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Week 12 or Final Visit..

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Weeks 4, 8 and 12 or Final Visit.
Change from baseline in fasting plasma glucose. | Weeks: 1, 2, 4, 8 and 12 or Final Visit.
Change from baseline in 1,5 anhydroglucitol. | Weeks 2, 4, 8 and 12 or Final Visit.
Change from baseline in proinsulin. | Weeks 4, 8 and 12 or Final Visit.
Change from baseline in insulin. | Weeks 4, 8 and 12 or Final Visit.
Change from baseline in proinsulin/insulin ratio. | Weeks 4, 8 and 12 or Final Visit.
Change from baseline in C-peptide. | Weeks 4, 8 and 12 or Final Visit.
Homeostasis model assessment insulin resistance. | Weeks 4, 8 and 12 or Final Visit.
Homeostasis model assessment beta-cell function. | Weeks 4, 8 and 12 or Final Visit.
Incidence of marked hyperglycemia (fasting plasma glucose ≥200 mg/dL [≥11.10 mmol/L]). | Weeks 1, 2, 4, 8 and 12 or Final Visit.
Incidence of rescue. | Weeks 1, 2, 4, 8 and 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin ≤6.5%. | Week 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin ≤7.0%. | Week 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin improvement ≥1.0%. | Week 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin improvement ≥1.5%. | Week 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin improvement ≥2.0%. | Week 12 or Final Visit.
Fasting lipids (triglycerides, total cholesterol, high-density lipoprotein and low-density lipoprotein cholesterol). | Weeks 4, 8, and 12 or Final Visit.
Postprandial area under the concentration-time curve and peak 2-hour values of plasma glucose, insulin and C-peptide during a 3-hour mixed-meal tolerance test in a subset of subjects. | Week 12 or Final Visit.
Plasma concentration of SYR-619. | Week 8.
Physical examination findings (including a clinical examination of skin and digits). | At All Visits
Vital sign measurements. | At All Visits
Body temperature measurements. | Week 12 or Final Visit.
12-lead electrocardiogram tracings. | Week 12 or Final Visit.
Incidence of adverse events. | At All Visits
Incidence of hypoglycemia (blood glucose <60 mg/dL [<3.33 mmol/L]) in the presence of symptoms or blood glucose <50 mg/dL [<2.78 mmol/L]) regardless of symptoms). | At All Visits
Clinical laboratory evaluations (hematology and serum chemistry). | At All Visits
Clinical laboratory evaluation (urinalysis). | Week 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda